CLINICAL TRIAL: NCT03682692
Title: ACEI/CCB Versus ACEI/DIU Combination Antihypertensive Therapy in Chinese Hypertensive Patients (ACvAD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACvAD
Record Dates: First submitted 2018-09-18; First posted 2018-09-25 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Randomization and treatment: Potentially eligible patients should receive a 24-hour ambulatory blood pressure monitoring measurement before randomization. After stratification by centers and whether receive antihypertensive treatment, eligible patients will be randomly divided into two groups, taking benazepril 10 mg/amlodipine besylate 5mg fixed-dose combination (1 tablet once a day) or benazepril 10 mg/hydrochlorothiazide 12.5 mg fixed-dose combination (1 tablet once a day). If the systolic/diastolic blood pressure higher than 140/90 mmHg during follow-up visits, the dosage can be increased to 2 tablets once a day. If the systolic/diastolic blood pressure still ≥140/90 mmHg, bisoprolol 5 mg (1 tablet once a day) or doxazosin controlled-release tablets 4 mg (1 tablet once a day) or spironolactone 20 mg (1 tablet once a day) can be added during the following follow-up visits.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACEI/CCB (Experimental)
  Interventions: Drug: ACEI/CCB
- ACEI/DIU (Experimental)
  Interventions: Drug: ACEI/DIU

INTERVENTIONS:
Drug: ACEI/CCB — benazepril 10 mg / amlodipine besylate 5 mg fixed-dose combination
  Arms: ACEI/CCB
Drug: ACEI/DIU — benazepril 10 mg / hydrochlorothiazide 12.5 mg fixed-dose combination
  Arms: ACEI/DIU

SUMMARY:
1. Study name: ACEI/CCB versus ACEI/DIU combination antihypertensive therapy in Chinese hypertensive patients (ACvAD)
2. Rationale:Most current hypertension guidelines recommend the combination therapy of an angiotensin-converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB) with a calcium antagonists (CCB) or thiazide diuretics (DIU). However, whether the two combination treatments have similar antihypertensive effects in Chinese hypertensive patients is still lack of clinical evidence, especially randomized controlled trials using ambulatory or home blood pressure measurement as the main evaluation method.
3. Study design: This study is a multi-center, randomized and controlled clinical trial with two equally sized treatment groups: ACEI/CCB group and ACEI/DIU group.
4. Study population: Men or women over 18 years (n=580) meeting the inclusion/exclusion criteria.
5. Randomization and treatment: Potentially eligible patients should receive a 24-hour ambulatory blood pressure monitoring measurement before randomization. After stratification by centers and whether receive antihypertensive treatment, eligible patients will be randomly divided into two groups, taking benazepril 10 mg/amlodipine besylate 5mg fixed-dose combination (1 tablet once a day) or benazepril 10 mg/hydrochlorothiazide 12.5 mg fixed-dose combination (1 tablet once a day).
6. Follow up: All patients should sign an informed consent form before entering the study. The follow-up period is 6 months.
7. Sample size estimation: a total of 580 patients should be enrolled in this study.

DETAILED DESCRIPTION:
1. Study name: ACEI/CCB versus ACEI/DIU combination antihypertensive therapy in Chinese hypertensive patients (ACvAD)
2. Medicine: Benazepril 10 mg/amlodipine besylate 5 mg fixed-dose combination, benazepril 10 mg/hydrochlorothiazide 12.5 mg fixed-dose combination.
3. Rationale: A meta-analysis of 42 studies showed that the combination of two antihypertensive drugs is better than monotherapy to control blood pressure. Most patients with grade 2 or higher hypertension need two or more antihypertensive drugs to control blood pressure. Antihypertensive therapy with fixed-dose combination can better control blood pressure and improve patient compliance, as well as reduce adverse effect. For untreated patients with high blood pressure level, the guidelines recommend that combination therapy can be used initially. The fixed-dose combination can control blood pressure to target, as well as improve patient compliance by reducing the number of tablets. Most current hypertension guidelines, including the Chinese guidelines for the management of hypertension, recommend the combination therapy of an angiotensin-converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB) with a calcium antagonists (CCB) or thiazide diuretics (DIU). However, whether the two combination treatments have similar antihypertensive effects in Chinese hypertensive patients is still lack of clinical evidence, especially randomized controlled trials using ambulatory or home blood pressure measurement as the main evaluation method. This randomized controlled clinical trial will be carried out in 580 Chinese hypertensive patients. By measuring office blood pressure, 24-hour ambulatory blood pressure and home blood pressure, the blood pressure lowering effect of benazepril 10 mg/amlodipine besylate 5 mg fixed-dose combination and benazepril 10 mg/hydrochlorothiazide 12.5 mg fixed-dose combination will be compared.
4. Objective: The primary objective is to evaluate the reduction of 24-hour ambulatory systolic blood pressure in the ACEI/CCB group compared with the ACEI/DIU group after 6 months of antihypertensive treatment. The secondary objectives are to compare the reduction of 24-hour, daytime, night-time, home and office systolic and diastolic blood pressure after 6 months of study medication treatment.
5. Study design: This study is a multi-center, randomized and controlled clinical trial with two equally sized treatment groups: ACEI/CCB group and ACEI/DIU group.
6. Study population: With the age over 18 years, newly diagnosed grade 1-2 hypertensive patients or grade 1-2 hypertensive patients with monotherapy whose blood pressure not controlled, having systolic blood pressure ranged from 140 to 179 mmHg or (and) diastolic blood pressure ranged from 90 to 109 mmHg, can enter a 4-week run-in period before randomization. During the run-in period, all patients take benazepril 10 mg daily, and have an office visit every two weeks. After taking benazepril for 4 weeks continually with no adverse effect, patients with the mean office blood pressure of the last two visits between 140 and 179 mmHg in systolic or (and) between 90 and 109 mmHg in diastolic are eligible for randomization. Eligible patients will switch to take study medication after randomization. A one-week home blood pressure measurement should be performed before randomization by using an automatic device. Exclusion criteria include: suspected or confirmed secondary hypertension; history of coronary heart disease, myocardial infarction, heart failure, stroke or dementia; other drugs that might affect blood pressure; serum levels of ALT, AST, TBL equal or higher than twice of the upper limit; serum creatinine ≥1.5 mg/dL (133 μmol/L); urine protein positive; serum potassium >5.5 mmol/L or <3.5 mmol/L; history of gout or serum uric acid ≥420 μmol/L for male or ≥360 μmol/L for female; elderly patients need caring; or patients who are participating other clinical trials.
7. Randomization and treatment: Potentially eligible patients should receive a 24-hour ambulatory blood pressure monitoring measurement before randomization. After stratification by centers and whether receive antihypertensive treatment, eligible patients will be randomly divided into two groups, taking benazepril 10 mg/amlodipine besylate 5 mg fixed-dose combination (1 tablet once a day) or benazepril 10 mg/hydrochlorothiazide 12.5 mg fixed-dose combination (1 tablet once a day). If the systolic/diastolic blood pressure higher than 140/90 mmHg during follow-up visits, the dosage can be increased to 2 tablets once a day. If the systolic/diastolic blood pressure still ≥140/90 mmHg, bisoprolol 5 mg (1 tablet once a day) or doxazosin controlled-release tablets 4 mg (1 tablet once a day) or spironolactone 20 mg (1 tablet once a day) can be added during the following follow-up visits.
8. Follow up: All patients should sign an informed consent form before entering the study. A validated Omron automatic device should be used to measure the sitting blood pressure in the clinic. Patients will be followed up every month with sitting office blood pressure measured and medical history recorded. Before each follow-up visit, a one-week home blood pressure measurement should be performed using an automatic Omron device; 24-hour ambulatory blood pressure monitoring, electrocardiogram, blood and urine biochemical tests should be repeated at the end of the 6 months of follow-up.
9. Sample size estimation: The primary outcome is the reduction of 24-hour ambulatory systolic blood pressure in the ACEI/CCB group compared with the ACEI/DIU group after 6 months of antihypertensive treatment. Assuming the difference between groups is 2.5 mmHg and the standard deviation is 10 mmHg, α is 0.05, and the power is 80%, the sample size of each group should be 252 patients. Accounting for 15% of add-up, each group needs 290 eligible patients. The total number of patietns is 580. The data will be analyzed by SAS software, and the t-test will be used to compare the continuous variables of two groups.
10. Timeline: Ethical review: November 2017; Enrollment: January 2018-June 2020; End of follow-up: December 2020. At the same, abstract of the main results will be submitted to domestic or international scientific conferences. The main results will be published in an international medical journal.
11. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
1. the age over 18 years,
2. newly diagnosed grade 1-2 hypertensive patients or grade 1-2 hypertensive patients with monotherapy whose blood pressure not controlled, having systolic blood pressure ranged from 140 to 179 mmHg or (and) diastolic blood pressure ranged from 90 to 109 mmHg,
3. can enter a 4-week run-in period before randomization. During the run-in period, all patients take benazepril 10 mg daily, and have an office visit every two weeks. After taking benazepril for 4 weeks continually with no adverse effect, patients with the mean office blood pressure of the last two visits between 140 and 179 mmHg in systolic or (and) between 90 and 109 mmHg in diastolic are eligible for randomization. Eligible patients will switch to take study medication after randomization. A one-week home blood pressure measurement should be performed before randomization by using an automatic device. Patient should agree to participate in the trial, and can pay follow-up visits.

Exclusion Criteria:

1. suspected or confirmed secondary hypertension
2. history of coronary heart disease, myocardial infarction, heart failure, stroke or dementia
3. other drugs that might affect blood pressure
4. serum levels of ALT, AST, TBL equal or higher than twice of the upper limit
5. serum creatinine ≥1.5 mg/dL (133 μmol/L)
6. urine protein positive
7. serum potassium >5.5 mmol/L or <3.5 mmol/L
8. history of gout or serum uric acid ≥420 μmol/L for male or ≥360 μmol/L for female
9. elderly patients need caring
10. patients who are participating other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
24-hour ambulatory systolic blood pressure reduction | 6 months
  the change of 24-hour ambulatory systolic blood pressure in the ACEI/CCB group compared with the ACEI/DIU group after 6 months of antihypertensive treatment

SECONDARY OUTCOMES:
reduction of other blood pressure measurements | 6 months
  the change of 24-hour, daytime, night-time, home and office systolic and diastolic blood pressure after 6 months of study medication treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

REFERENCES:
- [Derived] Huang QF, Zhang D, Luo Y, Hu K, Wu Q, Qiu H, Xu F, Wang ML, Chen X, Li Y, Wang JG; ACEI/CCB Versus ACEI/DIU Combination Antihypertensive Therapy in Chinese Hypertensive Patients (ACvAD) investigators. Comparison of two single-pill dual combination antihypertensive therapies in Chinese patients: a randomized, controlled trial. BMC Med. 2024 Jan 24;22(1):28. doi: 10.1186/s12916-023-03244-4. PMID 38263021